CLINICAL TRIAL: NCT00124085
Title: Asthma in a Decentralized Patient Population: Is Traditional Disease Management Enough? A Randomized, Controlled Trial Comparing Traditional Care to Two Systems of Disease Management for a Decentralized Population of Patients in South Texas
Brief Title: Asthma in a Decentralized Patient Population: Is Traditional Disease Management Enough?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: South Texas Veterans Health Care System (U.S. Federal Agency); Brooke Army Medical Center (U.S. Federal Agency); 59th Medical Wing (U.S. Federal Agency); TRICARE Southwest (Unknown); Department of Health and Human Services (U.S. Federal Agency); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 034-5001-057
Record Dates: First submitted 2005-07-22; First posted 2005-07-26 (Estimated); Last update posted 2012-08-09 (Estimated); Status verified 2012-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Disease Management

INTERVENTIONS:
Behavioral: Disease Management
Behavioral: Disease Management + Educational Home Visits

SUMMARY:
This is a health services demonstration project that evaluates three methods of health care delivery for the management of individuals with symptoms of asthma. This study will evaluate the impact of a telephonic asthma disease management process, with and without a home intervention program, on preventing asthma-related morbidity through patient/family asthma education.

The investigators' central thesis is that comprehensive clinical disease management protocols for the management of asthma will improve clinical outcomes; reduce fiscal resource consumption; and improve both patient satisfaction and patient quality of life. Additionally, individualized, in-home patient education and environmental assessment, when added to the telephonic protocol, will further improve these measures. However, incremental improvement will vary according to the population's access to care.

DETAILED DESCRIPTION:
This trial addresses the real-world concerns of asthma management through a disease management approach that will assist both the patient and the primary care physician by providing education, additional outpatient resources and additional access to health care personnel. This approach will stress empowering the patient to participate in his or her own health care at a higher level, which, in the case of asthma, is critical to wellness.

In a cooperative network of San Antonio medical centers, civilian and military, with a collective mission to care for military beneficiaries and the underserved patients of South Texas, this trial will evaluate the clinical benefits, as well as the cost savings, of a chronic disease management intervention in asthma. This study will fill a conspicuous gap in the medical literature by addressing the effectiveness of disease management through a large, decentralized, randomized, controlled trial.

DISEASE MANAGEMENT INTERVENTION

The project will use asthma disease management protocols and educational materials developed by the National Jewish Medical and Research Center. The program will be fully available in both English and Spanish, allowing a direct test of its impact on the State's vulnerable Hispanic population. Based on the principles of comprehensive disease management, National Jewish Medical and Research Center has developed a disease management program for asthma (DMP: Asthma) which addresses continuity of care by integrating traditional treatment methods with a program that focuses on creating a stronger partnership between the patient and the healthcare team, as well as greater patient empowerment. The primary program goal is empowering patients with the tools and resources they need for better self management of their prescribed treatment regimens and control of their environment. The program incorporates practice guidelines outlined by the National Heart, Lung, and Blood Institute (NHLBI) at the National Institutes of Health (NIH).

HOME VISIT INTERVENTION

In addition, the demonstration will evaluate the addition of a home-based disease management protocol focusing on patient education, to test for incremental improvement. Patients will be taught about their disease (symptoms, treatment, appropriate action plans), as well as about the healthcare system (how and when to access it). Based on the principles of comprehensive disease management and the unique needs of South Texas residents, the South Texas Asthma Management Program (STAMP) is designed for a diverse, mobile, underserved patient population. The protocol delivers up-front home-based education and environmental assessment, with follow-up visits focused on reinforcement of the earlier messages. The program ensures access to a primary care provider for patients who lack this critical member of the healthcare team. It also provides multiple resources for social services and guidance in appropriately accessing the healthcare system. The goal of the program is to equip patients, who have barriers to access due to a number of factors (lack of phone, language, remote location, etc), to navigate the healthcare system and effectively receive the care they need.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of asthma
* One or more of the following:

  * Acute visit with the primary diagnosis of asthma within the previous 6 months. (Includes visits to physician's office, emergency department, or any other health care facility.); OR
  * Three or more refills for inhaler medicine in the past 6 months, based on review of pharmaceutical records; OR
  * Diagnosis of asthma based on asthma symptoms and pulmonary function testing.

Exclusion Criteria:

* Other lung disease(s) with a possible reactive component (i.e. chronic obstructive pulmonary disease [COPD])
* Any diagnosis requiring chronic systemic steroids
* Enrollment in any other asthma disease management program
* Pregnancy
* Plan to reside at current residence for less than 12 months.

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1053
Dates: Start 2003-10; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Symptom-free days
Quality of Life Questionnaire (AQLQ, PAQLQ)
Rate of asthma-related hospitalizations over 18 months of enrollment
Rate of asthma-related emergency room (ER) visits over 18 months of enrollment

SECONDARY OUTCOMES:
Pulmonary function testing
SF-36
Days of school/work missed
Drug usage

CONTACTS AND LOCATIONS:
Overall Officials: Gregory L Freeman, MD, Principal Investigator — University of Texas; Jay I Peters, MD, Principal Investigator — University of Texas; Stephen Inscore, MD, Principal Investigator — University of Texas; Autumn Dawn Galbreath, MD, Study Director — University of Texas

REFERENCES:
- [Derived] Galbreath AD, Smith B, Wood PR, Inscore S, Forkner E, Vazquez M, Fallot A, Ellis R, Peters JI. Assessing the value of disease management: impact of 2 disease management strategies in an underserved asthma population. Ann Allergy Asthma Immunol. 2008 Dec;101(6):599-607. doi: 10.1016/S1081-1206(10)60222-0. PMID 19119703